CLINICAL TRIAL: NCT05045430
Title: Post Market Surveillance Study to Confirm the Ongoing Safety and Performance of Silver II Non-woven Dressing in Chronic and Acute Wounds
Brief Title: PMS Study to Confirm the Ongoing Safety and Performance of Silver II Non-woven Dressing in Chronic and Acute Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silver II Non-Woven 001
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Intervention (Experimental): Subjects will undergo treatment of their chronic or acute wound as indicated in the instructions for use with Silver II Non-Woven Dressing
  Interventions: Device: Silver II Non-Woven Dressing

INTERVENTIONS:
Device: Silver II Non-Woven Dressing — Assigned interventions Subjects will undergo treatment of their chronic and acute wounds as indicated in instructions for use with Silver II Non-Woven dressings.
  Subjects will be evaluated as follows:
  Full Patient and wound assessment, Informed consent. Wound Assessment, application of dressings, (At each scheduled dressing change.) Wound Assessment, removal of dressings, (At each scheduled dressing change.) The patients will be evaluated at each dressing change over six-week period (per Advanced Medical Solution Product) or until the wound is healed to extent that the use of Silver II Non-Woven dressing is no longer indicated from the time that the patient has been recruited.
  The assessment of the presence and reduction of the signs and symptoms of Infection.

SUMMARY:
Post Market Surveillance Study to confirm the safety and performance of Silver II Non-Woven Dressing in Chronic and Acute Wounds

DETAILED DESCRIPTION:
The design of the study is an open-label, multicentre, single arm clinical trial in subjects with moderate to heavily exuding infected chronic and acute wounds consisting of Pressure ulcers, Leg ulcers, Diabetic ulcers, Post-operative surgical wounds, Graft and donor sites, Cavity wounds, Trauma wounds (dermal lesions, trauma injuries or incisions) and Superficial and partial thickness burns. The performance data from this study will support clinically meaningful rates of successful improvement in the signs and symptoms of infection, without re-infection during 6-week treatment and follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 18 years or above. (Females must not be pregnant and if of reproductive age should be using contraception).
* Patients who are able to understand and give informed consent to take part in the study.
* Have one or more of the following: Pressure ulcer, Leg ulcer, Diabetic ulcers, Post-operative surgical wounds, Graft and donor sites, Cavity wounds, Trauma wounds (dermal lesions, trauma injuries or incisions) and superficial and partial thickness burn wounds that are infected, or are at high risk of infection , that are moderate to heavy levels of exudate.
* For Partial Thickness Second Degree Burns that require grafting - only those grafts with single thickness mesh grafts that have X % epithelialization will be enrolled [Note: % epithelization to be added once sites/countries are chosen as this is specific to the territory where the Silver II Non Woven Dressing study is likely to be performed].

Exclusion Criteria:

* Patients who are known to be non-compliant with medical treatment,
* Patients who are known to be sensitive to any of the device components
* Subject is pregnant or actively breastfeeding;
* Subject has a known sensitivity to Silver;
* Life expectancy of <6 months;
* Maximum burn area of > 20% total body area. Using the rule of nines assessment tool. [Note: criteria to be confirmed once sites/countries are chosen]
* Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the Silver II Non-Woven Dressing | No worsening of any signs/ symptoms of infection at 6 weeks or if infection resolved prior to 6 weeks, that no new evidence of infection occurred during the 6 week treatment follow up.
  Effectiveness (performance) of the Silver II Non-Woven Dressing will be evaluated for efficacy success according to the following success criteria:
  Reduction in signs and symptoms of infection from baseline as defined as
  The change from the Investigator's opinion of infection being present to no longer being present, or If the Investigator determines infection is still present there is improvement in severity of at least two.

SECONDARY OUTCOMES:
User satisfaction with the Silver II Non-Woven Dressing. | immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  To establish clinician and user satisfaction Clinician satisfaction with the device (conformability & ease of use) this will be assessed using a Likert type scale. (Very satisfied, Satisfied and not Satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Parthiban Vinayakam, Principal Investigator — Queen Elizabeth Queen Mother Hospital
Locations (8):
- Nianwi Healthcare, Germiston, South Africa
- United Kingdom (7):
  - Queen Elizabeth the Queen Mother Hospital, Margate, Kent
  - Castlegate and Derwent Surgery, Cockermouth
  - HMC Health, London
  - Nottingham University Hospitals City Hospital, Hucknall Rd,, Nottingham
  - University Hospitals Plymouth NHS Trust - Derriford Hospital, Plymouth
  - Berkshire Healthcare NHS Foundation 57-59 Bath Rd,, Reading
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: No